CLINICAL TRIAL: NCT03639064
Title: A Phase II, Randomized, Open-label, Double-blind, Two-center Study to Evaluate the Tolerability, Safety and Dose-finding of Oil Cannabis Preparation for Pain in Parkinson's Disease
Brief Title: Cannabis Oil for Pain in Parkinson's Disease
Acronym: MDC-CAN-PD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Collaborators: Parkinson Society Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 17-6086.0
Record Dates: First submitted 2018-07-04; First posted 2018-08-20 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2021-11

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — nabiximols

STUDY DESIGN:
Intervention Model Description: This is an interventional, phase II, randomized, open-label, double-blind, two-centre study to evaluate the safety, tolerability, and dose-finding of Cannabis oil preparation for pain in Parkinson's disease.
  Mixed oil cannabis preparation consisting of 3 differing formulations of ∆-9THC and CBD is clinically available in Canada as CanniMed®. The 3 differing formulations of CanniMed® oils contain varying proportions of ∆-9THC and CBD in the following ratios: 18:0; 10:10; 1:20. A total of 15 patients will be block randomized to one of the three groups. Each patient will receive one formulation of CanniMed® Oil only, with 5 patients per group.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This will be a double-blind study. The different cannabis oil formulations have the same colour, taste and smell. Study investigators will be blind to the dose/formulation of cannabis oil. Unblinding will only be performed in the event of a Serious AE. The site PI will maintain a randomization list kept in a locked secure 24h a day accessible location for emergency unblinding.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CanniMed® Oil 1:20 formulation (Experimental): ∆9-THC: 1.0 mg/mL; CBD: 20.0 mg/mL
  Interventions: Drug: Cannabis Oil
- CanniMed® Oil 10:10 formulation (Experimental): ∆9-THC: 9.8 mg/mL; CBD: 9.9 mg/mL
  Interventions: Drug: Cannabis Oil
- CanniMed® Oil 18:0 formulation (Experimental): ∆9-THC: 18.3 mg/mL; CBD: 0.2 mg/mL
  Interventions: Drug: Cannabis Oil

INTERVENTIONS:
Drug: Cannabis Oil — Mixed oil cannabis preparation consisting of 3 differing formulations of ∆-9THC and CBD is clinically available in Canada as CanniMed®. The 3 differing formulations of CanniMed® oils contain varying proportions of ∆-9THC and CBD in the following ratios: 18:0; 10:10; 1:20.
  All CanniMed® oil formulations consist of cannabinoids extracted from dried cannabis, and diluted in olive oil.

SUMMARY:
Full Title: A phase II, randomized, open-label, double-blind, two-center study to evaluate the tolerability, safety and dose-finding of oil cannabis preparation for pain in Parkinson's disease.

Short title: Cannabis oil for pain in Parkinson's disease Sample Size: N = 15 Study Population: Patients with Parkinson's disease and pain, without cognitive impairment.

Study Duration: July 2018 - July 2019

Study Agent/ Intervention: Cannabis oil: mixed oil cannabis preparation consisting of 3 different formulations of ∆-9THC and cannabidiol - 18:0; 10:10; and 1:20 respectively. Cannabis oil will be administered orally once per day, as required for pain; or taken 4h before bedtime, if no pain.

Primary objective: to determine the safety and tolerability of different formulations of Cannabis oil for pain in PD patients (incidence and severity of adverse events).

Secondary objective: to assess change from the start of treatment (V2) to end of treatment (V5) in frequency and severity of pain, sleep, dystonia and motor symptoms in PD patients.

DETAILED DESCRIPTION:
BACKGROUND AND RATIONALE Pain is a common symptom in PD and is reported in up to 50 % of patients. Pain in PD has been classified as musculoskeletal, dystonic (particularly in OFF-periods), radicular and central pain, and is frequently associated with muscle rigidity, postural abnormalities and bradykinesia. Often, the presence of pain in PD is associated with the daily fluctuations in the motor symptoms of PD. In addition, some patients experience 'off-dystonia' which affects the toes and feet, with painful cramps and posturing. The treatment of pain in PD patients with such fluctuating symptoms involves optimizing the dose of levodopa or other dopaminergic drugs to treat the OFF periods. Frequently, the pain does not resolve on altering the PD medication and remains difficult to treat.

Cannabis Sativa (marijuana) and its major psychoactive constituent, delta-9- tetrahydrocannabinol(Δ9THC) have been used for centuries to treat pain. The mechanism of action is likely mediated via cannabinoid receptors (CB1 and CB2) in basal ganglia and spinal circuits. Because of these potential therapeutic properties, several synthetic and naturally occurring cannabinoid preparations have been manufactured. Cannabinoids have been demonstrated to alleviate allodynia or hyperalgesia in animal models of pain; the effect on pain modulation may be secondary to CB1 receptors in the amygdala, thalamus, spinal cord and dorsal root ganglion. Several recent clinical studies have demonstrated the potential efficacy of synthetic and naturally occurring cannabinoids in pain. Synthetic cannabinoids such as nabilone and nabiximols are now licensed as add-on therapy in multiple sclerosis and advanced cancer for relief of pain. A Canadian systematic review of randomized clinical trials of cannabinoids (cannabis, nabilone, dronabinol and nabiximols) for the treatment of chronic non-cancer pain (neuropathic pain, mixed chronic pain, rheumatoid arthritis, fibromyalgia) concluded that cannabinoids are modestly effective. Other cannabinoids found in cannabis sativa include cannabidiol (CBD). CBD potentially lacks a psychoactive effect, and appears to act via non-CB receptor-mediated actions including ion channels and enzymes. Pre-clinical studies suggest anti-inflammatory, analgesic, anti-nausea, anti-emetic, anti-psychotic, anti-ischemic, anxiolytic, and anti-epileptiform actions. Thus, the advantage of CBD in PD is a potentially lesser risk of cognitive dysfunction and psychosis.

Currently, there is an oil preparation (CanniMed® Oil) in Canada, with the advantage of ease of administration. CanniMed® Oil is a mixed oil preparation that contains both Δ9THC and CBD, of varying proportions of Δ9THC (more psychoactive component) and CBD (18:0; 10:10; 1:20 respectively). Investigators of this study have experience in conducting trials using synthetic cannabinoids in movement disorders, including PD. Investigators have demonstrated tolerability, but limited efficacy, of short-term administration of clinically available oral tablet cannabinoids in idiopathic dystonia. More specifically in PD, investigators have assessed nabilone for the treatment of levodopa-induced dyskinesia with documented efficacy. Of interest to the current proposal, in this study, investigators also found an improvement in painful OFF-period limb dystonia in 2 out of 7 subjects. It is unknown if this effect is a specific analgesic effect or related with an anti-dystonia effect.

STUDY HYPOTHESIS Despite the major advances in understanding the pathophysiology of the endocannabinoid system, there are many unknowns in the use of cannabinoids for medical purposes. To date, clinical studies with cannabinoids in PD have been inconclusive and the use of cannabinoids remains controversial due to a lack of well-powered confirmatory clinical studies and obvious safety concerns. However, the known efficacy of cannabinoids in reducing pain suggests that PD-related pain may also be a reasonable target for cannabinoids. Combined with the potential rationale for reducing dystonia, we hypothesize that cannabinoids could reduce pain in PD, regardless of the PD-specific pain cause.

Primary Outcome

Safety:

* Incidence and severity of adverse events
* Maximum tolerated dose (MTD)

Tolerability:

* Ability to remain on assigned treatment
* Withdrawal rates due to adverse events

Secondary Outcomes: Assess change from baseline in the King's Parkinson Disease Pain scale (KPPS).

Other Outcomes: Assess change from baseline in frequency and severity of pain, sleep, dystonia and PD motor symptoms, using the following measurement tools:

* Visual Analogue Scale for Pain
* MDS-UPDRS part III
* UDysRS - Dystonia part 2 subscores
* Clinical Global Impression of pain severity (severity and improvement)
* Epworth Sleepiness Scale

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects;
* Aged >18y
* International Parkinson and Movement Disorder Society (MDS) Clinical Diagnostic Criteria for Parkinson Disease.
* Bothersome Pain - Defined as Severity score of 2 or more (Moderate pain of some distress to the patient); and Frequency score of 2 or more (at least 1 episode/week) in at least one pain domain according to King's Parkinson Disease Pain Scale (KPPS, see supplements);
* On stable PD medications in the month prior to enrollment.
* Drugs used to treat pain, including dopaminergic drugs, analgesics, non-steroidal anti-inflammatories and opiates will be allowed to be continued during the study period but doses must be unchanged.
* Women of childbearing age must be non-pregnant and using a reliable method of contraception and have a negative pregnancy test at screening. Acceptable methods of contraception include using oral injected or implanted methods of hormonal contraceptives for at least 3 months prior to randomization and the partner should also use a barrier method (e.g. condom) with spermicidal foam/gel/film/cream/suppository during this study. Additional pregnancy testing will be completed if necessary throughout the study duration.
* Subject agrees not to drive for the duration of the study.

Exclusion Criteria:

* Secondary parkinsonism (as per MDS Diagnostic Criteria).
* Previous serious adverse event or hypersensitivity to cannabis or cannabinoids
* Current use of cannabinoids or marijuana within 90 days prior to screening.
* Cognitive impairment or dementia (Montreal Cognitive Assessment/MoCA < 24).
* Current substance use disorder according to the Diagnostic and Statistical Manual of Mental Disorder Fifth Edition (DSM-5) and lifetime history of dependence on cannabis or diagnosis of cannabis use disorder (CUD) according to the DSM-5
* History of clinically significant impulse control disorders: QUIP-RS- part A-D ≥ 10 and part E ≥ 7.
* Current suicidal ideation within one year prior to the second Screening Visit as evidenced by answering "yes" to Questions 4 or 5 on the suicidal ideation portion of the C-SSRS or attempted suicide within the last 5 years.
* Symptomatic orthostatic hypotension or drop in (standing from sitting) blood pressure of >20 mmHg (systolic) and >10 mmHg (diastolic).
* Significant hepatic disease (AST, ALT, ALP >2xUpper Normal Limit).
* Normal renal function (defined as serum creatinine level <133 µmol/L and Estimated Glomerular Filtration Rate (eGFR) greater than or equal to 60)
* Uncontrolled and severe cardiovascular disease, as per clinical judgment.
* History of problematic substance abuse, or substance use disorder, whether of alcohol, prescription drugs or illicit drugs
* Other contra-indication as per Health Canada recommendation for use of cannabis - see reference 21.
* Inability or unwillingness of subject to give written informed consent.
* Participation in another investigational study at the time of recruitment or during the prior month.
* Clinical use of any exclusionary drugs listed in Appendix I of this protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) in each individual | From baseline (Visit 1) to end of study (Visit 5); total 35 days of intervention.
  MTD will be defined as the dose of each CanniMed® preparation for which the subject was able to be on for a minimum of 1 week, without the occurrence of an AE or suspected AE, with the severity grading of 2 or higher (CTCAE v.4.0)
Treatment-emergent adverse events (safety) | From baseline (Visit 1) to end of study (Visit 5); total 35 days of intervention.
  Determine the incidence and severity of adverse events by direct patient questioning, physical examination and ancillary testing as per protocol

SECONDARY OUTCOMES:
Collect the King's Parkinson Disease Pain scale (KPPS) scores in the intervention group, adjusted for baseline scores. | From baseline (Visit 1) to Follow-up phone call (1 week after Visit 5); Total 35 days
  KPPS is a validated, disease-specific scale with seven domains (different types of pain) including 14 items, each item scored by severity (0-3) multiplied by frequency (0-4) with a total possible score range from 0 to 168.

OTHER OUTCOMES:
Changes in the Visual Analogue Scale for Pain (adjusted for baseline scores) | From baseline (Visit 1) to end of study (Visit 5); total 35 days.
  The score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity.
Changes in the MDS-UPDRS part III (adjusted for baseline scores) | From baseline (Visit 1) to end of study (Visit 5); total 35 days.
  The score assesses the motor signs of PD and ranges between 0-137.
Changes in the UDysRS - Dystonia part 2 subscores (adjusted for baseline) | From baseline (Visit 1) to end of study (Visit 5); total 35 days.
  The scale is divided in 2 parts. Part 2A is administered by the rater (one question) and focuses on time spent with off-dystonia. Part 2B is a component of the Patient Questionnaire that covers three questions on the impact of painful off-dystonia on experiences of daily living. The score ranges between 0-16.
Changes in the Clinical global Impression of pain severity and improvement | From baseline (Visit 1) to end of study (Visit 5); total 35 days.
  The Clinical Global Impression - Severity scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. The Clinical Global Impression - Improvement scale (CGI-I) is a 7 point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention.
Changes in The Epworth Sleepiness Scale (ESS) (adjusted for baseline) | From baseline (Visit 1) to end of study (Visit 5); total 35 days.
  The ESS is a self-administered questionnaire with 8 questions. Respondents are asked to rate, on a 4-point scale (0-3), their usual chances of dozing off or falling asleep while engaged in eight different activities. The ESS score (the sum of 8 item scores, 0-3) can range from 0 to 24.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Fox, MD, PhD, Principal Investigator — UHN - Toronto Western Hospital - 399 Bathurst Street, McLaughlin pavilion, 7th Floor Toronto, ON, M5T 2S8 - Canada
Locations (2):
- Canada (2):
  - Parkinson's Disease and Movement Disorders Clinic - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Movement Disorders Clinic, Toronto Western Hospital, 399, Bathurst St, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Negre-Pages L, Regragui W, Bouhassira D, Grandjean H, Rascol O; DoPaMiP Study Group. Chronic pain in Parkinson's disease: the cross-sectional French DoPaMiP survey. Mov Disord. 2008 Jul 30;23(10):1361-9. doi: 10.1002/mds.22142. PMID 18546344
- [Result] Ha AD, Jankovic J. Pain in Parkinson's disease. Mov Disord. 2012 Apr;27(4):485-91. doi: 10.1002/mds.23959. Epub 2011 Sep 23. PMID 21953990
- [Result] More SV, Choi DK. Promising cannabinoid-based therapies for Parkinson's disease: motor symptoms to neuroprotection. Mol Neurodegener. 2015 Apr 8;10:17. doi: 10.1186/s13024-015-0012-0. PMID 25888232
- [Result] Fox SH, Henry B, Hill M, Crossman A, Brotchie J. Stimulation of cannabinoid receptors reduces levodopa-induced dyskinesia in the MPTP-lesioned nonhuman primate model of Parkinson's disease. Mov Disord. 2002 Nov;17(6):1180-7. doi: 10.1002/mds.10289. PMID 12465055
- [Result] Engler B, Freiman I, Urbanski M, Szabo B. Effects of exogenous and endogenous cannabinoids on GABAergic neurotransmission between the caudate-putamen and the globus pallidus in the mouse. J Pharmacol Exp Ther. 2006 Feb;316(2):608-17. doi: 10.1124/jpet.105.092718. Epub 2005 Oct 7. PMID 16214880
- [Result] Lynch ME, Ware MA. Cannabinoids for the Treatment of Chronic Non-Cancer Pain: An Updated Systematic Review of Randomized Controlled Trials. J Neuroimmune Pharmacol. 2015 Jun;10(2):293-301. doi: 10.1007/s11481-015-9600-6. Epub 2015 Mar 22. PMID 25796592
- [Result] Kluger B, Triolo P, Jones W, Jankovic J. The therapeutic potential of cannabinoids for movement disorders. Mov Disord. 2015 Mar;30(3):313-27. doi: 10.1002/mds.26142. Epub 2015 Feb 4. PMID 25649017
- [Result] Koppel BS, Brust JC, Fife T, Bronstein J, Youssof S, Gronseth G, Gloss D. Systematic review: efficacy and safety of medical marijuana in selected neurologic disorders [RETIRED]: report of the Guideline Development Subcommittee of the American Academy of Neurology. Neurology. 2014 Apr 29;82(17):1556-63. doi: 10.1212/WNL.0000000000000363. PMID 24778283
- See also: HealthCanada. Information for Health Care Professionals. Cannabis (marihuana, marijuana) and the cannabinoids — http://www.hc-sc.gc.ca/dhp-mps/alt_formats/pdf/marihuana/med/infoprof-eng.pdf